CLINICAL TRIAL: NCT00512785
Title: An Open-label Study to Evaluate the Long-term Safety and Efficacy of Imidafenacin in Patients With Overactive Bladder
Brief Title: Long-term Safety and Efficacy of Imidafenacin in Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRP197-T301/ONO-8025-12
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Overactive Bladder
Keywords: Imidafenacin; KRP-197/ONO-8025; overactive bladder; antimuscarinic
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — imidafenacin

ARMS (2):
- E1 (Experimental)
  Interventions: Drug: imidafenacin, KRP-197/ONO-8025
- E2 (Experimental)
  Interventions: Drug: imidafenacin, KRP-197/ONO-8025

INTERVENTIONS:
Drug: imidafenacin, KRP-197/ONO-8025 — 0.1 mg BID for 52 weeks
  Arms: E1
Drug: imidafenacin, KRP-197/ONO-8025 — 0.1 mg BID for 12 weeks and 0.2 mg BID for 52 weeks
  Arms: E2

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of imidafenacin.

ELIGIBILITY:
Inclusion Criteria:

* Men and Woman equal or > 20 years old
* Patients with urgency, urinary frequency and urgency incontinence

Exclusion Criteria:

* Patients with genuine stress incontinence
* Patients suffering from complications such as bladder tumor, urinary tract stone and symptomatic urinary tract infection
* Patients suffering from complications contraindicating the use of antimuscarinic medication
* Patients with polyuria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety Measures: adverse events, laboratory tests, 12-lead ECG, vital signs, post-void residual volume | 64 weeks

SECONDARY OUTCOMES:
Efficacy measures: number of urgency incontinence episodes per week, number of incontinence episodes per week, number of micturitions per day, number of urgency episodes per day, severity of urgency, urine volume voided per micturition, Quality of Life | 64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshifumi Hirahara, Study Director — Kyorin Pharmaceutical Co.,Ltd; Toshihiko Konomi, Study Chair — Ono Pharmaceutical Co. Ltd
Locations (2):
- Japan (2):
  - Kanto Region, Kanto
  - Kinki Region, Kinki